CLINICAL TRIAL: NCT04893876
Title: The OPERa Study: A Multicenter Observational Prospective Cohort Study to Evaluate Determinants of Long-Term Quality of Life Following Restorative Proctectomy for Rectal Cancer Treatment
Brief Title: The OPERa Study: Evaluating QoL After Rectal Cancer Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Associate Professor, Jewish General Hospital
Other Study IDs: MP-05-2021-2615
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer; Quality of Life; Bowel Dysfunction; Sexual Dysfunction; Urinary Dysfunction; Emotional Distress; Surgery
MeSH Terms: conditions — Rectal Neoplasms; Intestinal Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advances in rectal cancer management have significantly reduced morbidity and mortality. The most commonly performed operation for rectal cancer is restorative proctectomy (RP), leaving up to 70% with long-term bowel dysfunction called Low Anterior Resection Syndrome (LARS). LARS manifests as stool frequency, incontinence and difficult defecation. LARS, along with other functional impairments such as sexual and urinary dysfunction (SUD), can impact quality of life (QoL) and cause emotional distress. High-quality longitudinal data on these sequalae are lacking, leading to variable estimates of their prevalence, risk factors and prognosis. Most studies are European, cross-sectional, lack pre-treatment evaluation and long-term follow-up, and use inconsistent assessment measures. Thus, a North American study that evaluates patients longitudinally from diagnosis will provide quality data to fill this knowledge gap.

The main aim of the proposed study is to contribute evidence regarding the impact of LARS, SUD, emotional/financial distress, and patient activation on long-term post-treatment QoL in North American rectal cancer after RP.

This multicenter North American, observational, prospective cohort study relies on validated patient reported outcome measures (PROMs) at diagnosis, during and post-treatment. Patients from 20 sites will be recruited over 2 years and followed for 3 years. The primary endpoint is QoL as measured by the European Organization for Research & Treatment of Cancer QoL questionnaire. We anticipate accrual of 1200 patients. Factors associated with QoL will be explored. Impact of patient activation in relation to functional outcomes on QoL over time will be explored using a difference-in-differences approach. The study involves a multidisciplinary team who will provide expertise in research methodology, nursing, oncology and surgery.

The main contributions of this study are 1) provision of reference baseline North American values for important rectal cancer PROMs for clinical and research use, 2) an understanding of the evolution of functional outcomes and QoL post-treatment to counsel patients peri-operatively and throughout survivorship, and 3) to provide the basis for future tailored programs to support rectal cancer survivors.

DETAILED DESCRIPTION:
Advances in rectal cancer management have significantly reduced morbidity and mortality. The most commonly performed operation for rectal cancer is restorative proctectomy (RP), leaving up to 70% with long-term bowel dysfunction called Low Anterior Resection Syndrome (LARS). LARS manifests as stool frequency, incontinence and difficult defecation. LARS, along with other functional impairments such as sexual and urinary dysfunction (SUD), can impact quality of life (QoL) and cause emotional distress. There is no well-established treatment strategy for LARS or SUD. High-quality longitudinal data on these sequalae are lacking, leading to variable estimates of their prevalence, risk factors and prognosis. Most studies are European, cross-sectional, lack pre-treatment evaluation and long-term follow-up, and use inconsistent assessment measures. Thus, a North American study that evaluates patients longitudinally from diagnosis will provide quality data to fill this knowledge gap.

The main aim of the proposed study is to contribute evidence regarding the impact of LARS, SUD, emotional/financial distress, and patient activation on long-term post-treatment QoL in North American rectal cancer after RP. This study aims to address the following research questions: 1): How do North American rectal cancer patients who underwent RP experience changes in function (bowel, sexual and urinary), distress (emotional and financial) and QoL after RP from baseline through early and late timepoints following treatment? 2): How do patient-, disease-, treatment-, functional- and distress-related factors predict QoL at baseline and at early and late timepoints post-treatment?

This multicenter North American, observational, prospective cohort study relies on validated patient reported outcome measures (PROMs) at diagnosis, during and post-treatment. Patients from 20 sites will be recruited over 2 years and followed for 3 years. The primary endpoint is QoL as measured by the European Organization for Research & Treatment of Cancer QoL questionnaire. We anticipate accrual of 1200 patients. Estimating a 30% attrition rate, in 1000 different simulated datasets and α=0.05, we will be able to detect a 1 point difference in QoL 88% of the time (95%CI: 85.8, 90.0). Given that a 10-point difference is considered clinically significant, this sample size affords good precision. 1) QoL, LARS, SUD, emotional/financial distress will be measured at baseline, early (12 & 18 months) and late (2 & 3 years) timepoints. 2) Changes over time for each outcome will be studied using linear mixed models (LMM) and generalized LMM as appropriate to account for the hierarchical and longitudinal structure of the data. 3) Factors associated with QoL will be explored using LMM. 4) Impact of patient activation in relation to functional outcomes on QoL over time will be explored using a difference-in-differences approach. The study involves a multidisciplinary team who will provide expertise in research methodology, nursing, oncology and surgery.

The main contributions of this study are 1) provision of reference baseline North American values for important rectal cancer PROMs for clinical and research use, 2) an understanding of the evolution of functional outcomes and QoL post-treatment to counsel patients peri-operatively and throughout survivorship, and 3) to provide the basis for future tailored programs to support rectal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years with histopathologically confirmed adenocarcinoma of the rectum, defined as tumor ≤15cm from the anal verge who are planned for RP ± neoadjuvant treatment or WW (CRT alone without surgery).

Exclusion Criteria:

* Metastatic disease at diagnosis;
* Planned for abdominoperineal resection (APR), low Hartmann's or pelvic exenteration (PE);
* Cannot be contacted by telephone;
* Unable to read and comprehend English or French;
* Unable to give clear and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients >18 years with histopathologically confirmed primary rectal cancer ≤15cm from the anal verge who are planned for curative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Global Quality of Life (QoL) | 3 years
  Global QoL as measured by the European Organization for Research & Treatment of Cancer QoL questionnaire (EORTC QLQ-C30). Linear transformation is used to standardize raw score, so that scores range from 0 to 100; higher score represents better functioning or worse level of symptoms.

SECONDARY OUTCOMES:
Low Anterior Resection Syndrome Score | 3 years
  Measured by the Low Anterior Resection Syndrome Score (LARS Score). Score ranges from 0 to 42 points. 0-20: no LARS; 21-29 minor LARS; 30-42 major LARS.
Female Sexual Dysfunction | 3 years
  Measured for females by the Female Sexual Function Index (FSFI). FSFI: Minimum score 0, maximum score 36; higher score means better sexual function.
Male Sexual Dysfunction | 3 years
  Measured for males by the International Index of Erectile Function (IIEF). IIEF: Minimum score 0, maximum score 30. Higher score means better sexual function; higher score means better sexual function.
Female Urinary Dysfunction | 3 years
  Measured for females by the International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS). ICIQ-FLUTS: Minimum score 0, maximum score 48; Higher score means worse urinary symptoms.
Male Urinary Dysfunction | 3 years
  Measured for males by the International Prostate Symptom Score (IPSS). IPSS: Minimum score 0, maximum score 35. Higher sore means worse urinary symptoms.
Emotional Distress | 3 years
  Measured by the Hospital Anxiety and Depression Scale (HADS). HADS: Minimum score 0, maximum score 21; Higher score means greater emotional distress.
Financial Strain | 3 years
  Measured by a 7-level Likert scale questionnaire will be used to assess patients' perceived financial distress in relation to their disease. Minimum score 2, maximum score 14; Higher score means greater financial strain.
Patient Activation | 3 years
  Measured by the Patient Activation Measure (PAM-13). PAM-13: Minimum score 0, maximum score 100; increased score means greater patient activation.
Frailty | 3 years
  Measured by the Targeted Geriatric Assessment (TaGA). TaGA: Minimum score 0, maximum score 1; Higher score means increased frailty.

IPD SHARING:
Plan to Share IPD: No